CLINICAL TRIAL: NCT03924154
Title: A Phase 2a, Double-Blind, Placebo-Controlled Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Effects of RVT-1201 in Patients With Pulmonary Arterial Hypertension
Brief Title: A Study of RVT-1201 in Patients With Pulmonary Arterial Hypertension (ELEVATE 1)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to enroll
Sponsor: Altavant Sciences GmbH (Industry)
Collaborators: Altavant Sciences, Inc. (Unknown); PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RVT-1201-2001
Record Dates: First submitted 2019-04-05; First posted 2019-04-23 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2019-08

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary arterial hypertension (PAH); Pulmonary hypertension (PH); RVT-1201; Rodatristat ethyl; Tryptophan hydroxylase (TPH); Serotonin reduction; ELEVATE 1; KAR5417
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — rodatristat

STUDY DESIGN:
Intervention Model Description: Following screening assessments, PAH patients who meet all entrance criteria will be randomly assigned to receive one of the following treatments in a ratio of 2:1:
  * Arm 1 (n=24) - RVT-1201 Treatment: RVT-1201 immediate-release tablets will be administered orally, at a dose of 600 mg twice daily (BID), for a total of 6 weeks in addition to the patient's current standard of care (SOC) medication(s) for PAH.
  * Arm 2 (n=12) - Placebo Treatment: Matching placebo tablets will be administered orally, at a dose of 600 mg twice daily (BID), for a total of 6 weeks in addition to the patient's current SOC medication(s) for PAH.
  Participants will be followed in face-to-face visits with trial personnel every 2 weeks for 8 weeks (6 weeks of treatment plus a 2-week follow-up), with an additional phone call at Week 1, to assess drug effects and monitor safety during their treatments.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RVT-1201 (Experimental): RVT-1201 600 mg immediate-release tablet, administered orally twice daily with food for 6 weeks, in addition to the patient's current standard of care medication(s) for PAH (n=24 [Anticipated])
  Interventions: Drug: RVT-1201
- Placebo (Placebo Comparator): Matching placebo tablet, administered orally twice daily with food for 6 weeks, in addition to the patient's current standard of care medication(s) for PAH (n=12 [Anticipated])
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RVT-1201 — RVT-1201 600 mg immediate-release tablet
  Other Names: rodatristat ethyl
  Arms: RVT-1201
Drug: Placebo — Inactive pill manufactured to mimic RVT-1201 600 mg immediate-release tablet
  Other Names: Placebo (for RVT-1201)
  Arms: Placebo

SUMMARY:
This is an exploratory Phase 2a, randomized, double-blind, placebo-controlled, parallel-group, multicenter study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamic effects of RVT-1201 in patients with pulmonary arterial hypertension (PAH).

DETAILED DESCRIPTION:
This is an exploratory Phase 2a, randomized, double-blind, placebo-controlled, parallel-group, multicenter study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamic effects of RVT-1201 in patients with pulmonary arterial hypertension (PAH).

Study participation for each patient will last approximately 3 months and will consist of a screening period (up to 28 days in duration), a baseline period (day 1, pre-dose), a 6-week treatment period, and a 2-week follow-up period.

The study will enroll approximately 36 patients at approximately 20 centers across the United States and Canada.

ELIGIBILITY:
Key Inclusion Criteria:

* Symptomatic PAH belonging to one of the following types:

  * Idiopathic
  * Heritable
  * Drug- or toxin- induced
  * Associated with one of the following: connective tissue disease or congenital heart disease
* World Health Organization (WHO) Functional Class (FC) II or III
* PAH diagnosed by right heart cardiac catheterization prior to Screening
* Receiving standard of care treatment for PAH with oral monotherapy or dual therapy for at least 12 weeks prior to Screening at a dose which has been stable for at least 8 weeks prior to Screening
* If on a diuretic, dose must be stable for at least 4 weeks prior to Screening, with no changes anticipated during study participation
* 6-Minute Walk Distance (6MWD) between 150 and 500 meters at Screening and Baseline visits
* Plasma N-terminal pro B-type natriuretic peptide (NT-proBNP) level ≥ 300 pg/mL at Screening
* Ability and willingness to give written informed consent and to comply with the requirements of the study

Key Exclusion Criteria:

* PAH associated with human immunodeficiency virus (HIV) infection, portal hypertension or schistosomiasis
* Other types of pulmonary hypertension (PH):

  * Pulmonary hypertension due to left heart disease (WHO PH Group 2)
  * Pulmonary hypertension due to lung diseases and/or hypoxia (WHO PH Group 3)
  * Chronic thromboembolic pulmonary hypertension (WHO PH Group 4)
  * Pulmonary hypertension with unclear multifactorial mechanisms (WHO PH Group 5)
* Hospitalization for pulmonary hypertension within 12 weeks of screening
* Cardiopulmonary rehabilitation program based on exercise (planned, or started ≤ 12 weeks prior to Screening)
* Prostanoid or prostacyclin receptor agonist therapy within 12 weeks of screening
* Evidence of left-sided heart disease
* If Pulmonary function tests were done prior to screening, Pulmonary function tests demonstrate obstructive or restrictive lung disease
* Use of telotristat (Xermelo®) within the last 6 months
* Use of any investigational drug within 30 days or five half-lives (whichever is longer) prior to Screening, or 90 days if an investigational drug for PAH
* Have uncontrolled atrial fibrillation (AFib) or other uncontrolled arrhythmias
* Body mass index (BMI) >45 kg/m2
* Women of childbearing potential who are pregnant, planning to become pregnant, or lactating or female/male patients unwilling to use effective contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) and discontinuations due to AEs | 8 weeks
  Incidence of treatment-emergent adverse events (TEAEs), drug-related adverse events (AEs), and discontinuations due to AEs

SECONDARY OUTCOMES:
Concentration of biomarkers of serotonin biosynthesis in plasma | 8 weeks
  Absolute concentrations and percent change from baseline in plasma 5-hydroxyindoleacetic acid (5-HIAA) and plasma 5-hydroxytryptamine (5-HT, also known as serotonin) concentrations
Concentration of biomarkers of serotonin biosynthesis in urine | 8 weeks
  Concentration of urine 5-hydroxyindoleacetic acid (5-HIAA) will be normalized against urine creatinine concentration to determine absolute ratio and percent change from baseline in urine 5-HIAA:creatinine ratio
Study drug (RVT-1201) and active metabolite (KAR5417) plasma concentrations | 6 weeks
  Measured RVT-1201 and KAR5417 plasma concentrations from sparse sampling
Area under the plasma concentration versus time curve (AUC) of KAR5417 (the active metabolite of RVT-1201) | 6 weeks
  Measured KAR5417 plasma concentrations from sparse sampling will be used to assess the pharmacokinetic (PK) parameter AUC of KAR5417 administered twice daily in patients with PAH, by means of population PK (PopPK) analysis
Relationship between KAR5417 exposure and percent change from baseline in plasma concentrations of the serotonin-related biomarkers | 6 weeks
  Evaluate the relationship between exposure (area under the plasma concentration versus time curve [AUC]) of KAR5417 (the active metabolite of RVT-1201) and percent change from baseline in plasma concentrations of the serotonin-related biomarkers (5-HIAA and 5-HT)
Relationship between KAR5417 exposure and percent change from baseline in urine concentrations of the serotonin-related biomarkers | 6 weeks
  Evaluate the relationship between exposure (area under the plasma concentration versus time curve [AUC]) of KAR5417 (the active metabolite of RVT-1201) and percent change from baseline in urine 5-HIAA:creatinine concentration ratio

CONTACTS AND LOCATIONS:
Overall Officials: Ed Parsley, DO, Study Director — Altavant Sciences
Locations (23):
- United States (20):
  - Pulmonary Associates, PA, Phoenix, Arizona
  - University of California Davis Medical Center, Sacramento, California
  - SBPA Research LLC, Santa Barbara, California
  - University of Colorado, Aurora, Colorado
  - George Washington Medical Faculty Associates - Pulmonary Hypertension Program, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - Central Florida Pulmonary Group, P.A., Orlando, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Kentuckiana Pulmonary Research Center, Louisville, Kentucky
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Pulmonary Research Institute of Southeast Michigan, Farmington Hills, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Health Science Center at Houston, McGovern Medical School, Houston, Texas
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - London Health Sciences Centre, London, Ontario

IPD SHARING:
Plan to Share IPD: No